CLINICAL TRIAL: NCT01605461
Title: Metabolite Profile, Excretion Balance and Pharmacokinetics of BI 207127 NA Combined With [14C]-BI 207127 NA in Healthy Adult Male Volunteers After an 800 mg Single Oral Solution Dose; a Phase I, Single-arm, Open-label Trial
Brief Title: Study Evaluating Absorption, Distribution, Metabolism and Excretion (ADME) of Single Dose [14C]-BI 207127 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1241.22
Record Dates: First submitted 2012-05-09; First posted 2012-05-25 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Healthy

ARMS (1):
- BI 207127 NA (Experimental): Single oral solution dose of BI 207127 NA combined with [14C]-BI 207127 NA
  Interventions: Drug: BI 207127 NA

INTERVENTIONS:
Drug: BI 207127 NA — Single oral solution dose of BI 207127 NA combined with [14C]-BI 207127 NA

SUMMARY:
Phase 1 study to assess the pharmacokinetics and routes of elimination of a single oral dose of [14C]-BI 207127 and to characterize the metabolic profile following single dose administration.

ELIGIBILITY:
Inclusion criteria:

* Body mass index =18.5 and BMI = 29.9 kg/m2
* Subject is willing to avoid sun exposure from the first administration of the trial drug until the end of the study
* Male subjects must agree to minimise the risk of female partners becoming pregnant from the dosing day until three months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than three months prior to dosing or barrier contraception. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device, tubal ligation, or hormonal contraceptive for at least three months, or diaphragm with spermicide.
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria:

* Participation in more than one other radiolabelled investigational study drug trial within 12 months prior to check-in. The previous radiolabelled study drug must have been received more than 6 months prior to check-in for this study and the total exposure from this study and the previous study will be within the recommended levels considered safe, per 21 CFR 361.1 (eg. less than 5,000 mrem whole body annual exposure)
* Exposure to significant radiation (eg. serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to check-in
* Participation in another trial with an investigational drug within two months prior to administration of the trial drug or during the trial
* Use of drugs which might reasonably influence the results of the trial, including use of a broad spectrum antibiotic, within 10 days prior to administration of investigational medication in this trial or during the trial
* Intake of a drug with a half-life of >24 hours within the month prior to administration of trial medication, or if administration of trial medication would occur in the time period in which fewer than 10 half-lives had elapsed
* Surgery of the gastrointestinal tract (except appendectomy or cholecystectomy)
* Current smoker or smoker in last six months; alcohol abuse (more than 40 g/day); history of illicit drug abuse within the past 2 years
* Blood donation (more than 100 mL within four weeks prior to first administration of the trial drug or during the trial)
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms); a history of additional risk factors for torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* History of photosensitivity or recurrent rash
* Irregular defecation pattern (less than one bowel movement a day)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.22.001 Boehringer Ingelheim Investigational Site, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants received a single oral dose of 800 mg deleobuvir (BI 207127) sodium salt (NA) powder dissolved in a 20 mL solution of compendial grade sodium lauryl sulfate, tromethamine, polyethylene glycol 400, and water.
Period: Overall Study
Arm/Group | All Participants
Started | 12
Completed | 8
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who were dispensed study medication and were documented to have taken the dose of investigational treatment
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: AUC0-infinity of Plasma Deleobuvir
Description: Area under the plasma deleobuvir concentration-time curve over the time interval from 0 h extrapolated to infinity (AUC0-infinity)
Time Frame: 15 minutes (min) before drug administration and 30min, 1 hour (h), 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 15h, 24h, 36h, 48h, 72h and 96h after drug administration
Population: Pharmacokinetic analysis set (PK set) which included all subjects in the treated set who provided at least 1 observation for at least 1 primary PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | All Participants
Number analyzed (Participants) | 12
nmol*h/L | 19300 (56.5)

2. Primary Outcome: Cmax of Plasma Deleobuvir
Description: Maximum measured concentration (Cmax) of plasma deleobuvir
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | All Participants
Number analyzed (Participants) | 12
nmol/L | 3620 (54.2)

3. Primary Outcome: t1/2 of [14C]-Radioactivity in Plasma
Description: Terminal half life (T1/2) of [14C]-radioactivity in plasma
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | All Participants
Number analyzed (Participants) | 12
hours | 2.89 (36.4)

4. Primary Outcome: Excretion Balance of Total [14C]-Radioactivity
Description: Excretion balance of total [14C]-radioactivity (urine and faeces)
Time Frame: Before drug administration (24hours (h) to 15 minutes pre-dose) and 0h-24h, 24h-48h, 48h-72h, 72h-96h, 96h-120h, 120h-144h, 144h-168h, 168h-192h and 192h-216h after drug administration
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of radioactive dose recovered
Arm/Group | All Participants
Number analyzed (Participants) | 12
Percentage of radioactive dose recovered | 95.2 (1.29)

5. Primary Outcome: Excretion of Total [14C]-Radioactivity in Urine
Description: Excretion of total [14C]-radioactivity in urine
Time Frame: as for outcome 4
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of radioactive dose recovered
Arm/Group | All Participants
Number analyzed (Participants) | 12
Percentage of radioactive dose recovered | 0.137 (37.8)

6. Primary Outcome: Excretion of Total [14C]-Radioactivity in Faeces
Description: Excretion of total [14C]-radioactivity in faeces
Time Frame: as for outcome 4
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of radioactive dose recovered
Arm/Group | All Participants
Number analyzed (Participants) | 12
Percentage of radioactive dose recovered | 95.1 (1.29)

ADVERSE EVENTS:
Time Frame: From drug administration until end of study examination, up to 14 days
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vessel puncture site haemorrhage (General disorders) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.